CLINICAL TRIAL: NCT00214994
Title: A 12-Month, Open-Label, Flexible-Dosage Study to Evaluate the Safety and Efficacy of GABITRIL Treatment (up to 16 mg/Day) in Adults With Generalized Anxiety Disorder.
Brief Title: Study to Evaluate the Safety and Efficacy of GABITRIL Treatment in Adults With Generalized Anxiety Disorder.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C6671/3033/AX/US
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Tiagabine

INTERVENTIONS:
Drug: Gabitril

SUMMARY:
A 12-Month, Open-Label, Flexible-Dosage Study to Evaluate the Safety and Efficacy of GABITRIL Treatment in Adults with Generalized Anxiety Disorder.

ELIGIBILITY:
Subjects who have completed 10 weeks of double-blind treatment and the subsequent taper period in 1 of the 3 previous double-blind studies (studies C6671/3030/AX/US, C6671/3031/AX/US, or C6671/3032/AX/US).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2005-01; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Locations (93):
- United States (86):
  - Birmingham Research Group, Birmingham, Alabama
  - Pivotal Research Center, Mesa, Arizona
  - Pivotal Research, Peoria, Arizona
  - Southwestern Research, Beverly Hills, California
  - Valley Clinical Research, El Centro, California
  - Irvine Center for Clinical Res, Irvine, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pacific Institue for Medical, Los Angeles, California
  - Pharmacology Research Institute, Newport Beach, California
  - Pacific Clinical Research Medi, Orange, California
  - Pharmacology Research Institute, Riverside, California
  - Affiliated Research Institute, San Diego, California
  - HealthQuest Clinical Trials, San Diego, California
  - Clinical Innovations Inc., Santa Ana, California
  - Radiant Research Denver, Denver, Colorado
  - University of Connecticut, Farmington, Connecticut
  - University of Florida, Jacksonville, Florida
  - Miami Research Associates, Miami, Florida
  - Medicial Research Group of Central Florida, Orange City, Florida
  - Clinical Neuroscience Solution, Orlando, Florida
  - Roskamp Institute, Sarasota, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Clinical Neuroscience Solution, West Palm Beach, Florida
  - Atlanta Institue of Medicaine, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Carman Research, Smyrna, Georgia
  - Hawaii Clinical Research, Honolulu, Hawaii
  - American Medical Research, Aurora, Illinois
  - Cunningham Clinical Research, Edwardsville, Illinois
  - Henry Lahmeyer, MD, Northfield, Illinois
  - Midwest Center for Neurobehavi, Oakbrook Terrace, Illinois
  - Indiana University, Indianapolis, Indiana
  - Vince and Associates Clinical, Overland Park, Kansas
  - Hartford Research Ltd, Florence, Kentucky
  - Pedia Research, LLC, Owensboro, Kentucky
  - Four Rivers Clinical Research, Paducah, Kentucky
  - LSUHSC New Orleans, New Orleans, Louisiana
  - LSUHSC in Shreveport, Shreveport, Louisiana
  - Capital Clinical Research Asso, Rockville, Maryland
  - Dupont Clinical Research, Rockville, Maryland
  - University of Massachusetts, Worcester, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Summit Research Network Farmin, Farmington Hills, Michigan
  - Summit Research Network Michig, Okemos, Michigan
  - Regions Hospital, Saint Paul, Minnesota
  - Radiant Research Las Vegas, Las Vegas, Nevada
  - CNS Research Institute, Clementon, New Jersey
  - Center for Emotional Fitness, Moorestown, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Social Psychiatry Research Ins, Brooklyn, New York
  - Neurobehavioral Research, Inc., Lawrence, New York
  - Eastside Comprehensive Medical, New York, New York
  - Fieve Clinical Services, Inc., New York, New York
  - Medical and Behavioral, New York, New York
  - Medical Research Network, New York, New York
  - Behavioral Medical Research, Staten Island, New York
  - Medark Clinical Trials and Research, Morganton, North Carolina
  - Richard Weisler, MD and Assoc, Raleigh, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - North Coast Clinical Trials, Beechwood, Ohio
  - Hartford Research Group, Cincinnati, Ohio
  - Midwest Clinical Research Ctr, Dayton, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Pahl Pharmaceutical Research, Oklahoma City, Oklahoma
  - OCCI Eugene, Eugene, Oregon
  - Summit Research Network Inc., Portland, Oregon
  - OCCI, Inc., Salem, Oregon
  - Keystone Clinical Studies LLC, Norristown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - CNS Research Institute PC, Philadelphia, Pennsylvania
  - South East Health Consultants, Charleston, South Carolina
  - Carolina Clinical Research Ser, Columbia, South Carolina
  - Clinical Neuroscience Solution, Memphis, Tennessee
  - FutureSearch Trials, Austin, Texas
  - Claghorn-Lesem Research, Bellaire, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Fabre Research Clinics, Inc., Houston, Texas
  - R D Clinical Research, Lake Jackson, Texas
  - Croft Group Research Center, San Antonio, Texas
  - Radiant Research Salt Lake, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - Comprehensive Neuroscience Of, Arlington, Virginia
  - Northwest Clinical Research, Bellevue, Washington
  - Summit Seattle Boren, Seattle, Washington
  - Northbrook Research Center, Brown Deer, Wisconsin
  - Dean Foundation, Middleton, Wisconsin
- Canada (7):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - McMaster University Medical Ce, Hamilton, Ontario
  - Center for Addiction and Mental Health, Mood and Anxiety Program, Toronto, Ontario
  - Mood & Anxiety Disorders Ctr, Toronto, Ontario
  - Clinique Marie-Fitzbach, Québec, Quebec